CLINICAL TRIAL: NCT01024686
Title: Phase 1/2a Trial to Assess the Safety, Immunogenicity and Efficacy of Genetically-attenuated Plasmodium Falciparum Parasites p52-/p36- (GAP) Vaccine, Administered by Bite of Infected Anopheles Mosquito to Malaria-naïve Adults Living in the United States.
Brief Title: Phase 1/2a Trial of Pf GAP p52-/p36- Sporozoite Malaria Vaccine
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WR 1584
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-06

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- p52-p36- GAP Vaccine (Experimental): p52-/p56- GAP Vaccine: Administered by five bites from GAP-infected Anopheles mosquito.
  p52-/p56- GAP Vaccine: Administered by 200 bites from GAP-infected Anopheles mosquito.
  Challenge: Administered by five bites from Anopheles mosquitoes infected with wild type NF54 strain Plasmodium falciparum.
  Interventions: Biological: p52-/p36- GAP Vaccine; Biological: p52-p36- GAP Vaccine
- Infectivity Control (No Intervention): Active Control: Administered by five bites from Anopheles mosquitoes infected with wild type NF54 strain Plasmodium falciparum
- p52-p36- GAP Vaccine + Infectivity Challenge (Experimental): p52-/p36- GAP Vaccine: Five doses separated by 4-weeks, each administered by 200 bites from GAP-infected Anopheles mosquito.
  Challenge: Administered by five bites from Anopheles mosquitoes infected with wild type NF54 strain Plasmodium falciparum.
  Interventions: Biological: p52-/p36- GAP Vaccine

INTERVENTIONS:
Biological: p52-/p36- GAP Vaccine — Administered by five bites from GAP-infected Anopheles mosquito
  Arms: p52-p36- GAP Vaccine
Biological: p52-p36- GAP Vaccine — Administered by 200 bites from GAP-infected Anopeles mosquito
  Arms: p52-p36- GAP Vaccine
Biological: p52-/p36- GAP Vaccine — Five doses separated by 4-weeks, each administered by 200 bites from GAP-infected Anopheles mosquito
  Arms: p52-p36- GAP Vaccine + Infectivity Challenge

SUMMARY:
The purpose of this study is to assess safety and tolerability of escalating doses of a genetically attenuated parasite malaria vaccine (p52-/p36- GAP vaccine) in healthy malaria-naive adults. The study will also assess preliminary efficacy of p52-/p36- GAP vaccine following primary experimental challenge with P. falciparum sporozoites. Lastly, the study will assess immunogenicity of p52-/p36- GAP in malaria-naïve healthy adults and preliminary efficacy of p52-/p36- GAP vaccine following primary experimental re-challenge with P. falciparum sporozoites.

ELIGIBILITY:
Inclusion Criteria:

* A male or non-pregnant, non-lactating female 18 to 50 years of age (inclusive) at the time of enrollment
* Free of significant health problems as established by medical history, laboratory assessment and clinical examination before entering into the study
* Volunteers must have low cardiac risk factors according to the NHANES I criteria and a non-significant electrocardiogram (EKG) as determined by a expert consultant cardiologist
* Available to participate for duration of study
* Reproductive status: a female participant must:
* not be of reproductive potential: i.e. be surgically, medically or physiologically sterile, or
* if engages in sexual activity that could lead to pregnancy:
* agrees to consistently use contraception until 2 months after the last protocol visit. Contraception is defined as using 1 of the following methods:
* condoms (male or female) with or without a spermicide
* diaphragm or cervical cap with spermicide
* intrauterine device (IUD)
* hormonal contraception
* If the volunteer indicates he/she is active duty military (on the DCT sign-in page and intake form), approval from their supervisor through the Division Director using the Statement of Supervisor's Approval Form must be signed and on file prior to receipt of any test product
* Written informed consent must be obtained from the subject before screening procedures
* Prior to entry into this study, subjects must score at least 80% correct on a 10- question multiple-choice quiz that assesses their understanding of this study.

Exclusion Criteria:

* Prior receipt of any investigational malaria vaccine
* Use of any investigational or non-registered drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period
* Administration of any vaccine within 30 days of first study vaccination Any past history of malaria
* Planned travel to malarious areas during the study period
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* A family history of congenital or hereditary immunodeficiency
* Moderate or high 5-year cardiovascular risk as determined by NHANES 1 model
* An abnormal 12-lead electrocardiogram (EKG) suggestive of cardiac disease as determined by a clinician
* Seropositive for HIV, Hepatitis C virus (antibodies to HCV) and/or HBsAg
* Hepatomegaly, right upper quadrant abdominal pain or tenderness
* History of splenectomy
* Chronic or active neurologic disease including seizure disorder and chronic migraine headaches
* History of psoriasis and porphyria
* Acute or chronic, clinically significant pulmonary, cardiovascular, ocular, hematologic, hepatic or renal functional abnormality, as determined by physical examination or abnormal baseline laboratory screening tests and medical history review
* Administration of chronic (defined as more than 14 days) immunosuppressants or other immune-modifying drugs within six months of vaccination. For corticosteroids, this is defined as prednisone, or equivalent, 0.5 mg/kg/day. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period
* Current chronic use of medications known to cause drug reactions with chloroquine and/or atovaquone/proguanil such as cimetidine and metoclopramide.
* Current chronic use or use within one month prior to enrollment of antibiotics with anti-malarial effects such as tetracyclines for acne, sulfa drugs for recurrent urinary tract infections, etc.
* Pregnant or lactating female
* Female who is willing or intends to become pregnant during the study and for two (2) months after study completion
* Any history of allergic reaction or anaphylaxis to previous vaccination
* History of severe reactions to mosquito bites.
* Inability to make follow-up visits or complete diary cards
* Suspected or known current alcohol abuse/drug abuse as obtained by history and physical examination
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michele Spring, M.D., Principal Investigator — Walter Reed Army Institute of Research (WRAIR)
Locations (1):
- Walter Reed Army Institute of Research, Silver Spring, Maryland, United States

REFERENCES:
- [Result] Spring M, Murphy J, Nielsen R, Dowler M, Bennett JW, Zarling S, Williams J, de la Vega P, Ware L, Komisar J, Polhemus M, Richie TL, Epstein J, Tamminga C, Chuang I, Richie N, O'Neil M, Heppner DG, Healer J, O'Neill M, Smithers H, Finney OC, Mikolajczak SA, Wang R, Cowman A, Ockenhouse C, Krzych U, Kappe SH. First-in-human evaluation of genetically attenuated Plasmodium falciparum sporozoites administered by bite of Anopheles mosquitoes to adult volunteers. Vaccine. 2013 Oct 9;31(43):4975-83. doi: 10.1016/j.vaccine.2013.08.007. Epub 2013 Sep 8. PMID 24029408
- See also: First-in-human evaluation of genetically attenuated Plasmodium falciparum sporozoites administered by bite of Anopheles mosquitoes to adult volunteers. — https://www.ncbi.nlm.nih.gov/pubmed/24029408

RESULTS

PARTICIPANT FLOW:
Groups:
- p52-p36- GAP Vaccine: p52-/p36- GAP Vaccine: Administered by five bites from GAP-infected Anopheles mosquito.
  p52-p36- GAP Vaccine: Administered by 200 bites from GAP-infected Anopheles mosquito.
  Challenge: Administered by five bites from Anopheles mosquitoes infected with wild type NF54 strain Plasmodium falciparum.
- p52-p36- GAP Vaccine + Infectivity Challenge: p52-/p36- GAP Vaccine: Five doses separated by 4-weeks, each administered by 200 bites from GAP-infected Anopheles mosquito
  Challenge: Administered by five bites from Anopheles mosquitoes infected with wild type NF54 strain Plasmodium falciparum.
Period: Overall Study
Arm/Group | p52-p36- GAP Vaccine | Infectivity Control | p52-p36- GAP Vaccine + Infectivity Challenge
Started | 6 (July 11, 2010: unexpected adverse event, (1) participant) | 0 | 0
Completed | 6 | 0 ((0) participants because the clinical trial was terminated prior to enrollment.) | 0 ((0) participants because the clinical trial was terminated prior to enrollment.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No data is available for Infectivity Control or p52-p36- GAP Vaccine + Infectivity Challenge because the clinical trial was terminated prior to enrollment.
Groups:
- Total: Total of all reporting groups
Arm/Group | p52-p36- GAP Vaccine | Infectivity Control | p52-p36- GAP Vaccine + Infectivity Challenge | Total
Number analyzed (Participants) | 6 | 0 | 0 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 |  |  | 1
  Between 18 and 65 years | 5 |  |  | 5
  >=65 years | 0 |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  |  | 3
  Male | 3 |  |  | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Solicited Adverse Events (AE)
Time Frame: From administration of study vaccine through 7 days (± 1 days) post dosing
Population: (0) Zero participants analyzed because the study was terminated prior to enrollment.
Measure: Number; unit: events
Groups:
- p52-p36- GAP Vaccine: p52-/p36- GAP Vaccine: Administered by five bites from GAP-infected Anopheles mosquito
  p52-p36- GAP Vaccine: Administered by 200 bites from GAP-infected Anopheles mosquito
Arm/Group | p52-p36- GAP Vaccine | Infectivity Control | p52-p36- GAP Vaccine + Infectivity Challenge
Number analyzed (Participants) | 6 | 0 | 0
events | 52 |  |

2. Primary Outcome: Occurrence of Unsolicited AEs
Time Frame: From administration of study vaccine through 28 days (± 4 days) post dosing
Population: (0) Participants because clinical study was terminated before enrollment for Infectivity Control and p52-p36- GAP Vaccine + Infectivity Challenge.
Measure: Number; unit: events
Arm/Group | p52-p36- GAP Vaccine | Infectivity Control | p52-p36- GAP Vaccine + Infectivity Challenge
Number analyzed (Participants) | 6 | 0 | 0
events | 13 |  |

3. Primary Outcome: Occurrence of Laboratory Adverse Events (AE)
Description: Volunteers with any laboratory abnormality.
Time Frame: From administration of study vaccine through 7 days (± 1 days) post dosing
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | p52-p36- GAP Vaccine | Infectivity Control | p52-p36- GAP Vaccine + Infectivity Challenge
Number analyzed (Participants) | 6 | 0 | 0
Participants | 2 |  |

4. Primary Outcome: Detection of Breakthrough Peripheral Parasitemia by Thick Blood Film
Time Frame: From 7 days after administration of vaccine through 28 days (+ 4 days) post-dosing
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | p52-p36- GAP Vaccine | Infectivity Control | p52-p36- GAP Vaccine + Infectivity Challenge
Number analyzed (Participants) | 6 | 0 | 0
participants | 1 |  |

5. Primary Outcome: Occurrence of Serious Adverse Events (SAE)
Time Frame: baseline through 28 days
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | p52-p36- GAP Vaccine | Infectivity Control | p52-p36- GAP Vaccine + Infectivity Challenge
Number analyzed (Participants) | 6 | 0 | 0
participants | 1 |  |

6. Secondary Outcome: Development of Parasitemia and Time to Parasitemia After Primary Malaria Challenge Following Administration of GAP
Time Frame: From administration of study vaccine through the duration of the trial
Population: (0) Participants because clinical study was terminated before enrollment for primary malaria challenge
Arm/Group | p52-p36- GAP Vaccine | Infectivity Control | p52-p36- GAP Vaccine + Infectivity Challenge
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Development of Parasitemia and Time to Parasitemia After Re-challenge Following Administration of GAP
Time Frame: From administration of study vaccine through the duration of the trial
Population: (0) Participants because clinical study was terminated before enrollment for primary malaria challenge.
Arm/Group | p52-p36- GAP Vaccine | Infectivity Control | p52-p36- GAP Vaccine + Infectivity Challenge
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: P. Falciparum Specific Cell-mediated Immune Responses
Time Frame: From administration of study vaccine through the duration of the trial
Population: (0) data available because the clinical trial was terminated before DAY 90 blood draw for P. falciparum specific cell-mediated immune responses.
Arm/Group | p52-p36- GAP Vaccine | Infectivity Control | p52-p36- GAP Vaccine + Infectivity Challenge
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Description: This clinical study was withdrawn before enrollment of participants for arm 2 and arm 3. Therefore, no participants were at risk for adverse events from these arms.
Arm/Group | p52-p36- GAP Vaccine | Infectivity Control | p52-p36- GAP Vaccine + Infectivity Challenge
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | p52-p36- GAP Vaccine (N=6) | Infectivity Control (N=0) | p52-p36- GAP Vaccine + Infectivity Challenge (N=0)
Peripheral parasitemia (Infections and infestations) | 1 (1) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | p52-p36- GAP Vaccine (N=6) | Infectivity Control (N=0) | p52-p36- GAP Vaccine + Infectivity Challenge (N=0)
Fatigue (General disorders) | 4 (10) | NA | NA
Arthralgia (General disorders) | 3 (4) | NA | NA
Diarrhea (General disorders) | 1 (3) | NA | NA
Fever (General disorders) | 1 (1) | NA | NA
Malaise (General disorders) | 2 (6) | NA | NA
Myalgia (General disorders) | 3 (7) | NA | NA
Nausea/vomiting (General disorders) | 4 (13) | NA | NA
Headache (General disorders) | 6 (27) | NA | NA
Edema (Skin and subcutaneous tissue disorders) | 5 (8) | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 6 (19) | NA | NA
Induration (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA
Pain (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA
Puritus (Skin and subcutaneous tissue disorders) | 6 (18) | NA | NA
Anaemia (Blood and lymphatic system disorders) | 1 (1) | NA | NA
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | NA | NA
Otitis externa (Ear and labyrinth disorders) | 1 (1) | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 (1) | NA | NA
Toothache (Gastrointestinal disorders) | 1 (1) | NA | NA
Application site papules (General disorders) | 1 (1) | NA | NA
Feeling cold (General disorders) | 1 (1) | NA | NA
Feeling hot (General disorders) | 2 (3) | NA | NA
Injection site discoloration (General disorders) | 1 (1) | NA | NA
Injection site erythema (General disorders) | 2 (2) | NA | NA
Vaccination site pruritus (General disorders) | 1 (1) | NA | NA
Seasonal Allergy (Immune system disorders) | 1 (1) | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | NA | NA
Dizziness (Nervous system disorders) | 2 (6) | NA | NA
Insomnia (Nervous system disorders) | 1 (2) | NA | NA
Photophobia (Nervous system disorders) | 1 (1) | NA | NA
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (2) | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA
Rash papuar (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA
Scab (Skin and subcutaneous tissue disorders) | 1 (1) | NA | NA
Haemoglobin decreased (Investigations) | 2 (2) | NA | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | NA | NA
Confusion (Injury, poisoning and procedural complications) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No